CLINICAL TRIAL: NCT07253220
Title: Prospective, Randomized, Controlled Clinical Study Comparing TAF Monotherapy Versus ETV Combined With TAF on the Efficacy and Prognosis of Immunotherapy for Hepatitis B-Related Hepatocellular Carcinoma
Brief Title: TAF Monotherapy Versus ETV Combined With TAF on the Efficacy and Prognosis of Immunotherapy for Hepatitis B-Related Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, Ph.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: II2025-364-02
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis B; Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF Monotherapy (Other): TAF monotherapy (TAF 25mg qd)
  Interventions: Drug: TAF monotherapy
- ETV Combined with TAF (Other): ETV combined with TAF (ETV 0.5 mg qd +TAF 25 mg qd）
  Interventions: Drug: The arm will receive combination therapy (entecavir 0.5 mg once daily plus TAF 25 mg once daily); after HBV DNA becomes undetectable, the combination group will switch to TAF monotherapy.

INTERVENTIONS:
Drug: The arm will receive combination therapy (entecavir 0.5 mg once daily plus TAF 25 mg once daily); after HBV DNA becomes undetectable, the combination group will switch to TAF monotherapy. — Combination therapy (entecavir 0.5 mg once daily plus TAF 25 mg once daily)
  Arms: ETV Combined with TAF
Drug: TAF monotherapy — TAF monotherapy (TAF 25 mg once daily)
  Arms: TAF Monotherapy

SUMMARY:
Study Objective: To compare the efficacy and prognosis of systemic cancer therapy between TAF monotherapy and ETV plus TAF combination therapy in patients with unresectable, advanced hepatitis-B-related hepatocellular carcinoma (HBV-HCC).

Study Design: Prospective, interventional cohort study. Participants: Patients with histologically or radiologically confirmed unresectable, advanced HBV-HCC who are scheduled to receive immune-based systemic therapy at The Third Affiliated Hospital of Sun Yat-sen University. Detailed inclusion/exclusion criteria are provided below.

Intervention: Enrolled participants will be assigned to receive either TAF monotherapy or ETV combined with TAF for HBV suppression.

Primary Outcome: Overall survival (OS) at 24 months after initiation of systemic therapy, compared between the two HBV-treatment strategies.

Secondary Outcomes: Decline in HBV DNA and HBsAg levels at 1, 3, 12 and 24 months.

Sample Size: 120 HCC patients (60 per arm). Statistical Analysis: All analyses will be performed with SPSS. Continuous variables will be tested for normality (Shapiro-Wilk). Normally distributed data are presented as mean ± SD; non-normally distributed data as median (IQR). Twenty-four-month OS will be estimated by Kaplan-Meier curves and compared with a Cox proportional-hazards model adjusted for age, BCLC stage, AFP level, and ICI regimen. PFS will be compared using the log-rank test; ORR and HBV DNA undetectable rate will be compared with χ² tests. Inverse-probability-of-treatment weighting (IPTW) will address selection bias, and multiple imputation will handle missing data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, positive HBsAg for ≥ 6 months, and HBV DNA ≥ 2,000 IU/mL within 2 weeks before enrollment;

  * Histologically or clinically confirmed unresectable or metastatic hepatocellular carcinoma, Child-Pugh class A or B, ECOG performance status 0-1, and scheduled to receive systemic immunotherapy in the Department of Infectious Diseases, The Third Affiliated Hospital of Sun Yat-sen University;

    * At least one measurable lesion that has either not undergone local therapy or has progressed after local therapy, as defined by modified RECIST (mRECIST); ④ Estimated life expectancy ≥ 12 weeks; ⑤ Signed informed consent form for study participation

Exclusion Criteria:

* Co-infection with HCV or HIV; ② History of organ transplantation; ③ Presence of cardiac or renal insufficiency, or active autoimmune disease that constitutes a contraindication to immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
24-month overall survival (OS) after initiation of systemic therapy between TAF monotherapy and ETV plus TAF combination therapy in patients with unresectable, advanced HBV-related hepatocellular carcinoma. | 24 months
  24-month overall survival (OS)

IPD SHARING:
Plan to Share IPD: No